CLINICAL TRIAL: NCT04268758
Title: A Single-center Study Designed to Evaluate the Safety and Efficacy of a New Hygienic Device, Tulipon, in Adult Females With Normal Monthly Menstruation
Brief Title: A Single-center Study Designed to Evaluate the Safety and Efficacy of Tulipon
Status: Withdrawn | Type: Observational
Why Stopped: logistic and financial issues.
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Gals Bio Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: Tulipon-HMO-CTIL
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2020-04

CONDITIONS: Safety Issues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: tulipon — Tulipon is a new kind of hygienic device, used to collect the secreted menses during the bleeding phase of the menstruation.

SUMMARY:
Subjects who normally use tampons will use Tulipon device during one menstrual cycle. Baseline and post usage clinical evaluation will be performed for safety testing.

DETAILED DESCRIPTION:
Subjects use Tulipon device during one menstrual cycle. Baseline and post usage clinical evaluation will be performed for safety testing.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-45 years
2. Regular menstrual cycles (21-35 days)
3. Uses tampons every month for the last 2 months to handle their monthly bleeding.
4. Active Bleeding lasts at least 3 days
5. Willing not to change their feminine care or hygiene practices during their participation in the study (except as directed by the protocol and instructions for participants)
6. Non-pregnant, with no intentions to get pregnant during the clinical trial
7. Willing to use pads provided thought the study only for the duration of this study
8. Subject is able to comply with all the requirements of the study and agrees to participate in all the activities of the study
9. Signed written informed consent form (ICF) to participate in the study

Exclusion Criteria:

1. Pregnant or lactating women
2. Gave birth less than a 12 month prior to the study.
3. Virgin
4. Using medications to manage pain during active bleeding
5. Using intrauterine device or intrauterine device with hormones (Mirena)
6. Had experienced Toxic shock syndrome (TSS)
7. Previous diagnosis of primary or secondary dysmenorrhea
8. Previous diagnosis of endometriosis
9. Experiences urinary incontinence
10. Suffers from uterus or urine prolapse
11. Abnormal findings following the gynecological exam
12. Subjects with a known or suspected sensitivity to any of the device materials (Polyethylene, Polyurethane, Nylon, Cotton)
13. Been through a vaginal operation in the last 6 months prior to the study.
14. Participation in current or recent clinical trial within 30 days prior to baseline visit

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — women only.
Study Population: Adult females with normal monthly menstruation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
safety and efficacy of the Tulipon. | 1 month
  We will take vaginal cultures to show no vaginal infection. By questionnaire we will find out about leakage of period blood from the Tulipon.

IPD SHARING:
Plan to Share IPD: Undecided